CLINICAL TRIAL: NCT00559910
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of Once-Daily Orally Administered PH-797804 (0.5, 3, 6 And 10 MG) In Adults With Moderate To Severe Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: A Phase II, Study To Evaluate The Efficacy And Safety Of PH-797804 In Adults With Moderate To Severe Chronic Obstructive Pulmonary Disease (COPD).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6631011
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — PH 797804

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PH-797804 (Experimental): PH-797804 at four dose levels
  Interventions: Drug: PH-797804
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PH-797804 — PH-797804 at four dose levels
  Arms: PH-797804
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
PH-797804 is a potent ant-inflammatory drug that may reduce the inflammation that is associated with COPD. PH-797804 will be dosed to patients with COPD to evaluate its potential safety and efficacy profile in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including, the ages of 40 and 80 years.
* Subjects with a diagnosis, for at least 6 months, of moderate to severe COPD (GOLD) and who meet the criteria for Stage II-III disease, subjects must have had stable disease for at least 1 month prior to screening.
* Subjects must have a smoking history of at least 10 pack-years and be current smokers or ex-smokers that gave up > 6 months ago.

Exclusion Criteria:

* More than 2 exacerbations of COPD requiring treatment with oral steroids in the preceding year or hospitalization for the treatment of COPD within 3 months of screening or more than twice during the preceding year.
* History or presence of significant cardiovascular disease.
* ECG abnormalities.
* Significant concomitant clinical disease that could interfere with the conduct, safety or interpretation of results of this study.
* Evidence of organ or blood disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measures (AEs, 12-lead ECG, lab safety) during 6 weeks of treatment and up to 2 weeks post treatment. | 6 weeks
Spirometry measures during 6 weeks of treatment and up to 2 weeks post treatment. | 6 weeks

SECONDARY OUTCOMES:
Peak expiratory flow rate. | 6 weeks
Blood sample for pharmacogenomics | 6 weeks
Blood sample for pharmacokinetics | 6 weeks
Rescue bronchodilator usage. | 6 weeks
Dyspnea index scores. | 6 weeks
Global impression of change (patient and clinician). | 6 weeks
Symptom scores. | 6 weeks
Blood sample for biomarkers | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- Argentina (4):
  - Pfizer Investigational Site, La Plata, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires F.D.
  - Pfizer Investigational Site, Ciudad Autonoma de Buenos Aires (caba), Buenos Aires F.D.
  - Pfizer Investigational Site, Rosario, Santa Fe Province
- Australia (3):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Daw Park, South Australia
  - Pfizer Investigational Site, Nedlands, Western Australia
- Canada (5):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, Sainte-Foy, Quebec
- Chile (3):
  - Pfizer Investigational Site, Valparaíso, Región de Valparaíso
  - Pfizer Investigational Site, Providencia, Santiago, RM
  - Pfizer Investigational Site, Talca
- Czechia (6):
  - Pfizer Investigational Site, Cvikov
  - Pfizer Investigational Site, Kutná Hora
  - Pfizer Investigational Site, Liberec
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Strakonice
  - Pfizer Investigational Site, Tábor
- France (4):
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Perpignan
- Greece (3):
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Heraklion
  - Pfizer Investigational Site, Larissa
- Hungary (4):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Deszk
  - Pfizer Investigational Site, Pécs
  - Pfizer Investigational Site, Szombathely
- Netherlands (2):
  - Pfizer Investigational Site, Almere Stad
  - Pfizer Investigational Site, Zutphen
- Pfizer Investigational Site, Yaroslavl, Russia
- South Africa (3):
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Durban
- South Korea (2):
  - Pfizer Investigational Site, Anyang
  - Pfizer Investigational Site, Seoul
- Pfizer Investigational Site, Edinburgh, United Kingdom

REFERENCES:
- [Derived] MacNee W, Allan RJ, Jones I, De Salvo MC, Tan LF. Efficacy and safety of the oral p38 inhibitor PH-797804 in chronic obstructive pulmonary disease: a randomised clinical trial. Thorax. 2013 Aug;68(8):738-45. doi: 10.1136/thoraxjnl-2012-202744. Epub 2013 Mar 28. PMID 23539534
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631011